CLINICAL TRIAL: NCT02756637
Title: Neutrophil-to-Lymphocyte Ratio in Bladder Cancer: A Secondary Biomarker Analysis of SWOG 8710
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 15816
Record Dates: First submitted 2016-04-20; First posted 2016-04-29 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prognostic: Patients with NLR who completed curative therapy (surgery with or without chemo)
- Predictive: Patients with NLR who were assigned to a trial arm (chemo or no chemo)

SUMMARY:
The purpose of this study is to perform a secondary analysis of SWOG 8710 to assess NLRs value as a biomarker. Specifically, the investigators test two hypotheses: 1) that baseline NLR is correlated with overall survival after curative treatment for BC and 2) that baseline NLR is correlated with the survival benefit of NAC. The study will look at the data from participants of the SWOG 8710 study.

ELIGIBILITY:
Inclusion Criteria:

1. SWOG 8710 original trial inclusion criteria included:

   * Node-negative, muscle-invasive transitional cell carcinoma of the bladder, T2-T4aN0M0 per the AJCC 4th edition staging manual.
   * SWOG performance status of 0 or 1
   * Adequate organ function by lab criteria (WBC > 4,000 cells/mm3, platelets >150,000 cells/mm3, creatinine <1.5 md/dL (men) or <1.3 md/dL (women), baseline liver tests < 2 times normal limits)
2. Inclusion criteria for this secondary analysis are:

   * Eligible for original SWOG 8710 trial
   * Had complete blood count with differential prior to first treatment (radical cystectomy or NAC).

Exclusion Criteria:

1. SWOG 8710 original trial exclusion criteria included:

   * No age restrictions
   * Previous or concomitant malignancy other than bladder cancer or basal cell skin cancer
   * Prior pelvic radiation
   * Metastatic or incurable disease
   * Laboratory values exceeding those detailed in 3.1.c
2. Exclusion criteria for this secondary analysis are:

   * Ineligibility for the original SWOG 8710 study
   * Lack of complete blood count with differential prior to first treatment (cystectomy or NAC).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in SWOG 8710
Sampling Method: Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Christodouleas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prognostic Cohort: Patients with NLR who completed curative therapy (surgery with or without chemo)
- Predictive Cohort: Patients with NLR who were assigned to a trial arm (chemo or no chemo)
Period: Overall Study
Arm/Group | Prognostic Cohort | Predictive Cohort
Started | 317 | 317
Eligible for SWOG 8710 | 307 | 307
Had NLR Value | 263 | 263
Completed Curative Treatment | 230 | 0
Completed | 230 | 263
Not Completed | 87 | 54
Not completed — Not eligible for initial SWOG study | 10 | 10
Not completed — No available NLR value | 44 | 44
Not completed — Did not complete curative therapy | 33 | 0

BASELINE CHARACTERISTICS:
Population: Prognostic Cohort: Eligible for SWOG 8710, had NLR and completed curative treatment Predicitive Cohort: Eligible for SWOG 8710, had NLR and were assigned to a trial arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prognostic Cohort | Predictive Cohort | Total
Number analyzed (Participants) | 230 | 263 | 493
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 148 | 277
  >=65 years | 101 | 115 | 216
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 95
  Male | 185 | 213 | 398
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 230 | 263 | 493

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of participants who survived at 26 years are reported.
Time Frame: 26 years
Measure: Number; unit: participants
Arm/Group | Prognostic Cohort | Predictive Cohort
Number analyzed (Participants) | 230 | 263
participants | 58 | 58
Statistical Analysis 1: Comparison: Prognostic Cohort; The Hazard Ration is the ratio of survival rates between patients with high NLR and low NLR; Test type: Other; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.98 to 1.11]
Statistical Analysis 2: Comparison: Predictive Cohort; The Hazard Ration is the ratio of survival rates between patients with high NLR and low NLR; Test type: Other; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.90 to 1.14]

ADVERSE EVENTS:
Arm/Group | Prognostic Cohort | Predictive Cohort
Serious Adverse Events (participants affected / at risk) | 0/230 | 0/263
Other Adverse Events (participants affected / at risk) | 0/230 | 0/263

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes